CLINICAL TRIAL: NCT05230498
Title: Comparison of an Anatomy-based Fitting and a Conventional Fitting in Newly Implanted Cochlear Patients. Prospective Monocentric Randomized Double-blind Crossover Study.
Brief Title: Study of Sound and Speech Perception in New Cochlear Implanted Subjects Using or Not an Anatomy-based Fitting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: MEDEL_anatfit_Bordeaux_study
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Sensorineural Hearing Loss, Bilateral
Keywords: cochlear implant strategy; anatomy-based fitting
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: Two arms A and B:
  Arm A: patient's fitting with default fitting --> 6 weeks use --> tests and patient's fitting with anatomy-based fitting --> 6 weeks use --> tests Arm B: patient's fitting with anatomy-based fitting --> 6 weeks use --> tests and patient's fitting with default fitting --> 6 weeks use --> tests
Who Masked: Participant, Investigator
Masking Description: Double blind study: the patient and the investigator don't know the fitting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cochlear Implant (CI) with default fitting then anatomy-based fitting (Active Comparator): Cochlear Implant with default fitting first during 6 weeks then with anatomy-based fitting during 6 weeks
  Interventions: Device: default fitting then anatomy-based fitting
- Cochlear Implant (CI) with anatomy-based fitting then default fitting (Active Comparator): Cochlear Implant with anatomy-based fitting during 6 weeks then with default fitting during 6 weeks
  Interventions: Device: anatomy-based fitting then default fitting

INTERVENTIONS:
Device: anatomy-based fitting then default fitting — Cochlear implant with anatomy-based fitting then default fitting
  Arms: Cochlear Implant (CI) with anatomy-based fitting then default fitting
Device: default fitting then anatomy-based fitting — Cochlear implant with anatomy-based fitting then default fitting
  Arms: Cochlear Implant (CI) with default fitting then anatomy-based fitting

SUMMARY:
Main objective:

Compare the recognition of environmental sounds with an anatomy-based fitting and with a default fitting adult patients newly implanted with a MED-EL cochlear implant.

Secondary objectives:

Compare speech recognition in quiet with an anatomy-based fitting and with a default fitting in adult patients newly implanted with a MED-EL cochlear implant.

Compare speech recognition in noise with an anatomy-based fitting and with a default fitting in adult patients newly implanted with a MED-EL cochlear implant.

DETAILED DESCRIPTION:
Introduction: Cochlear implantation allows the rehabilitation of profound bilateral deafness, restoring speech perception and verbal communication when the traditional hearing aid no longer provides satisfactory hearing gain. A cochlear implant includes an electrode array and its functioning is based on the principle of cochlear tonotopy: each electrode encodes a frequency spectrum according to its position in the cochlea (high frequencies are assigned to the basal electrodes and low frequencies to the apical electrodes). The cochlear implant thus breaks down the frequency spectrum into a number of frequency bands via bandpass filters corresponding to the number of electrodes in the implant. During the fitting these bands can be modified by the audiologist. The fitting software developed by the manufacturers proposed a default fitting with a lower limit between 100 and 250 Hz according to the brands and an upper limit of about 8500 Hz. The frequency bands assigned to each electrode follow a logarithmic scale with the high frequencies for the basal electrodes and the low frequencies for the apical electrodes. This distribution takes into account the number of active electrodes but does not take into account the anatomy and the natural cochlear tonotopy specific to each patient. Several studies have analyzed the anatomical variations of the cochlear dimensions: size of the cochlea and the ratio between the contact surfaces of the electrodes with the cochlea are variable from one patient to another. The insertion depth during surgery is also variable due to parameters related to the patients as well as to the operator, which seems to impact the understanding of speech in noise. Mathematical algorithms have recently been developed to estimate the cochlear tonotopy of each patient from a CT scan assessment. CT imaging of the implanted ear combined with 3D reconstruction software, provides cochlear length measurements Using this approach it is possible to measure the position of each electrode relative to the cochlear apex. Recently, MED-EL (Austria) has developed a new approach based on CT-scan and tuning of the frequencies associated with each electrode using anatomical information of position of the electrodes in the cochlea: this fitting is called anatomy-based fitting.

Main objective:

Compare the recognition of environmental sounds with an anatomy-based fitting and with a default fitting adult patients newly implanted with a MED-EL cochlear implant.

Secondary objectives:

Compare speech recognition in quiet with an anatomy-based fitting and with a default fitting in adult patients newly implanted with a MED-EL cochlear implant.

Compare speech recognition in noise with an anatomy-based fitting and with a default fitting in adult patients newly implanted with a MED-EL cochlear implant.

Plan of the study:

It is a prospective open monocentric randomized crossover study: measures will be done on the patient at 6 weeks and 12 weeks post-activation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>= 18 years old) speaking French
* Patient who fulfils the criteria for cochlear implantation

Exclusion Criteria:

* retro-cochlear pathology: auditory neuropathy, vestibular schwannoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Recognition of Environmental sounds | at 6 weeks post-activation
  The environmental sound recognition is evaluated with the Environmental Sound Identification Test (TISE, Treville-Protain et al. 2019). The patient has to recognize 24 environmental sounds. Each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%).
Recognition of Environmental sounds | at 12 weeks post-activation
  The environmental sound recognition is evaluated with the Environmental Sound Identification Test (TISE, Treville-Protain et al. 2019). The patient has to recognize 24 environmental sounds. Each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%).

SECONDARY OUTCOMES:
Speech recognition in quiet | at 6 weeks post-activation
  The speech recognition in quiet is evaluated with 3 lists of 10 disyllabic words. The patient has to recognize 30 words. Each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%).
Speech recognition in quiet | at 12 weeks post-activation
  The speech recognition in quiet is evaluated with 3 lists of 10 disyllabic words. The patient has to recognize 30 words. Each good answer is scored 1 yielding a total between 0 and 1 (or 0% and 100%).
Speech recognition in noise | at 6 weeks post-activation
  The speech recognition in noise is evaluated with the French-language "Rapid speech in noise" (VRB) test (Leclerc et al. 2018). The speech level is at 65 dB SPL. The patient has to recognize 3 target words by sentence. The 8 sentences are played with signal-to-noise ratios between +18 dB and -3 dB by steps of 3 dB. The SRT50 (threshold for 50% intelligibility in noise) is obtained by SRT50 = 19,5 - R, with R = number of correct answers (on 24).
Speech recognition in noise | at 12 weeks post-activation
  The speech recognition in noise is evaluated with the French-language VRB test (Leclerc et al. 2018). The speech level is at 65 dB SPL. The patient has to recognize 3 target words by sentence. The 8 sentences are played with signal-to-noise ratios between +18 dB and -3 dB by steps of 3 dB. The SRT50 (threshold for 50% intelligibility in noise) is obtained by SRT50 = 19,5 - R, with R=number of correct answers (on 24).

CONTACTS AND LOCATIONS:
Overall Officials: Damien Bonnard, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No